CLINICAL TRIAL: NCT01543230
Title: Ceramic on Metal Total Hip System, CoMplete™ Acetabular Hip System
Brief Title: CoMplete™ Acetabular Hip System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew PMA
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09014
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Non-inflammatory Degenerative Joint Disease; Osteoarthritis; Post-traumatic Arthritis
Keywords: Non-Inflammatory Degenerative Joint Disease
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CoMplete™ Acetabular Hip System (CoM) (Experimental): Total hip arthroplasty (THA) using CoMplete™ Acetabular Hip System
  Interventions: Device: Total hip replacement

INTERVENTIONS:
Device: Total hip replacement — Total hip arthroplasty (THA) using CoMplete™ Acetabular Hip System

SUMMARY:
The primary objective of this investigation is to evaluate survivorship at ten years. For this post approval study (PAS), a maximum acceptable hazard of revision is assumed to be a constant 1% per year.

DETAILED DESCRIPTION:
This is a retrospective and prospective, non-randomized study of the Ceramic on Metal(CoM) device. This study will follow each subject through 10 years postoperatively. A total of 250 subjects will be enrolled in the investigation comprised of approximately 150 new PAS subjects and approximately 100 subjects recruited from the investigational device exemption study to the PAS.

ELIGIBILITY:
Inclusion Criteria:

* 1. If the subject:

  1. Was previously enrolled in the CoM IDE study with the Ceramic-on- Metal device, or
  2. Qualifies based on the approved labeling for the device; and
* 2. Is willing and able to provide informed patient consent for participation in the PAS study; and
* 3. Is willing and able to return for follow-up as specified by the PAS study protocol; and
* 4. Is willing and able to complete the hip outcomes questionnaire as specified by the PAS study protocol. A patient will be considered a "Valid Study Subject" when he/she has

  * consented to participate,
  * authorized release of Personal Health Information (PHI),
  * met all eligibility criteria through the operative stage, and
  * received the implant as noted in this protocol.

Exclusion Criteria:

* Subjects will be excluded if, in the opinion of the investigator, the subject does not qualify based on approved labeling requirements or Subject Inclusion criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Survivorship | 10 years
  Subjects will be seen each year through year 5 postoperatively for radiographic and clinical follow-up, and then at 8 and 10 years postoperatively for radiographic and clinical follow-up. Survivorship means the removal of either or both of the components (ceramic head or metal liner).

SECONDARY OUTCOMES:
Metal Ion Levels | 5 years, 8 years, and 10 years postoperatively
  A subset of subjects will be measured for serum cobalt, serum chromium, erythrocytes cobalt, erythrocytes chromium, whole blood cobalt, and whole blood chromium levels. These subjects will also be measured for BUN and creatine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Whalen, BS, DC, Study Director — DePuy Orthopaedics
Locations (6):
- United States (6):
  - Hip and Knee Arkansas Foundation, Little Rock, Arkansas
  - Orthopaedic Specialty Institute, Orange, California
  - Fort Collins, Colorado
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Seattle, Washington